CLINICAL TRIAL: NCT00087347
Title: An NCI-Sponsored Exploratory Study For Determining Optimum Timing For The Imaging Of Intravenous Superparamagnetic Particle Ferumoxytol (Code7228) For The Differentiation of Metastatic and Non Metastatic Lymph Nodes in Patients With Known Primary Cancer Scheduled For Possible Surgical Lymph Node Biopsy/Dissection
Brief Title: Magnetic Resonance Imaging of Lymph Nodes Using Ferumoxytol in Patients With Primary Prostate or Breast Cancer
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mukesh Harisinghani, MD, Associate Professor, Massachusetts General Hospital
Other Study IDs: CDR0000374491; MGH-2004-P-000681/2; NCI-6809
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Ferrosoferric Oxide; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Drug: ferumoxytol
Procedure: magnetic resonance imaging

SUMMARY:
RATIONALE: Diagnostic procedures such as magnetic resonance imaging (MRI) using ferumoxytol may improve the ability to detect cancer that has spread to the lymph nodes and may help plan effective cancer treatment.

PURPOSE: This clinical trial is studying how well MRI using ferumoxytol works in detecting metastases to the lymph nodes in patients with primary prostate cancer or primary breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the range of optimal timing for magnetic resonance imaging of lymph nodes after administration of ferumoxytol, in terms of assessing signal intensity using pre-defined pulse sequences in regions of interest and visual criteria, in patients with primary prostate or breast cancer who are scheduled to undergo surgical lymph node dissection or sampling.

Secondary

* Correlate MRI signal intensity with histological findings in patients undergoing this procedure.

OUTLINE: This is an open-label, pilot study.

Patients undergo a baseline MRI. Within 24 hours after the baseline MRI, patients receive ferumoxytol IV over 10-15 seconds (or over 1 hour). Patients then undergo MRI immediately after ferumoxytol administration (at the discretion of the principal investigator) and then at 24-28 hours.

Patients are followed at 2 weeks.

PROJECTED ACCRUAL: A total of 10-14 patients (6-8 with prostate cancer and 4-6 with breast cancer) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary prostate or breast cancer
* Suspected lymph node metastatic disease by standard MRI or CT scan
* Scheduled for surgical lymph node dissection or sampling
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* No prior ferritin > 800 ng/mL
* No prior transferrin saturation > 60%
* No history of iron overload or hemachromatosis

  * Patients with a clinical history of suspected iron overload or hemachromatosis must have normal serum iron, ferritin, and transferrin saturation

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* SGOT ≤ 2 times ULN

Renal

* Not specified

Other

* No requirement for monitored anesthesia during MRI
* No known allergic or hypersensitivity reaction to any of the following parenterally-administered preparations:

  * Iron
  * Dextran
  * Iron dextran
  * Iron polysaccharide
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for at least 1 month before and during study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior therapy for metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2004-09; Primary Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mukesh Harisinghani, MD, Study Chair — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Harisinghani M, Ross RW, Guimaraes AR, Weissleder R. Utility of a new bolus-injectable nanoparticle for clinical cancer staging. Neoplasia. 2007 Dec;9(12):1160-5. doi: 10.1593/neo.07940. PMID 18084623